CLINICAL TRIAL: NCT03523520
Title: Methylnaltrexone Versus Naloxegol in the Treatment of Opioid-Induced Constipation in the Emergency Department
Brief Title: Methylnaltrexone vs Naloxegol in the Treatment of Opioid-Induced Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Kara B. Goddard, PharmD, BCPS, Clinical Pharmacy Specialist, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011409 HS
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Constipation Drug Induced
Keywords: constipation; opioid
MeSH Terms: conditions — Constipation | interventions — methylnaltrexone; Tablets; naloxegol

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three groups i. Methylnaltrexone oral tablets (total 450 mg) + subcutaneous water injection ii. Methylnaltrexone 12mg subcutaneous injection + placebo sugar tablets iii. Naloxegol oral tablets (total 25 mg) + subcutaneous water injection
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each participant will be receiving one injection and tablets which have been randomly assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Methylnaltrexone oral tablets (Active Comparator): Methylnaltrexone oral tablets (total 450 mg) + subcutaneous water injection
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Interventions: Drug: Methylnaltrexone Bromide 150 mg Oral Tablet
- Methylnaltrexone subcutaneous injection (Active Comparator): Methylnaltrexone 12mg subcutaneous injection + sugar placebo tablet
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Interventions: Drug: Methylnaltrexone Bromide 12 MG/0.6 ML Subcutaneous Solution [RELISTOR]_#1
- Naloxegol oral tablets (Active Comparator): Naloxegol oral tablets (total 25 mg) + subcutaneous water injection
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Interventions: Drug: Naloxegol 25 MG Oral Tablet

INTERVENTIONS:
Drug: Methylnaltrexone Bromide 150 mg Oral Tablet — Methylnaltrexone Bromide 150 mg Oral Tablet
  Other Names: Relistor
  Arms: Methylnaltrexone oral tablets
Drug: Methylnaltrexone Bromide 12 MG/0.6 ML Subcutaneous Solution [RELISTOR]_#1 — Methylnaltrexone Bromide 12 MG Subcutaneous Solution
  Other Names: Relistor
  Arms: Methylnaltrexone subcutaneous injection
Drug: Naloxegol 25 MG Oral Tablet — Naloxegol 25 MG Oral Tablet
  Other Names: Movantik
  Arms: Naloxegol oral tablets

SUMMARY:
The purpose of this study is to compare the efficacy of subcutaneous versus oral mu-opioid receptor antagonist therapy in opioid induced constipation that is refractory to other bowel regimens.

DETAILED DESCRIPTION:
Opioid-induced constipation can lead to serious complications, including small bowel obstruction, fecal impaction, and bowel perforation. Not only are the medical complications potentially severe, patient quality of life can also be impacted. Two agents are currently available for opioid-induced constipation - oral and subcutaneous methylnaltrexone and oral naloxegol. Mechanistically, both agents antagonize the peripheral mu-opioid receptor in the gastrointestinal tract to decrease constipation without reversing the systemic analgesic effects of opiates. The literature currently available has evaluated the effectiveness of each agent, not the comparative effectiveness of these agents.

ELIGIBILITY:
Inclusion Criteria:

* Complaint of opioid-induced constipation refractory to other therapy (enemas, laxatives, stool softeners)
* Age≥18y/o
* Not pregnant or lactating (negative urinary pregnancy test)
* No contraindication to Methylnaltrexone or Naloxegol

Exclusion Criteria:

* Age<18y/o
* Pregnancy or lactation
* Contraindication to Methylnaltrexone or Naloxegol
* Assigned NPO
* Small bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KARA B GODDARD, PharmD, BCPS, Principal Investigator — UNIVERSITY OF MISSOURI HEALTH CARE
Locations (1):
- Kara B. Goddard, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowers BL, Crannage AJ. The Evolving Role of Long-Term Pharmacotherapy for Opioid-Induced Constipation in Patients Being Treated for Noncancer Pain. J Pharm Pract. 2019 Oct;32(5):558-567. doi: 10.1177/0897190017745395. Epub 2017 Dec 5. PMID 29207909
- [Result] Jones R, Prommer E, Backstedt D. Naloxegol: A Novel Therapy in the Management of Opioid-Induced Constipation. Am J Hosp Palliat Care. 2016 Nov;33(9):875-880. doi: 10.1177/1049909115593937. Epub 2015 Jul 6. PMID 26150678
- [Result] Anantharamu T, Sharma S, Gupta AK, Dahiya N, Singh Brashier DB, Sharma AK. Naloxegol: First oral peripherally acting mu opioid receptor antagonists for opioid-induced constipation. J Pharmacol Pharmacother. 2015 Jul-Sep;6(3):188-92. doi: 10.4103/0976-500X.162015. PMID 26312011

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylnaltrexone Oral Tablets: Methylnaltrexone oral tablets (total 450 mg)
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Methylnaltrexone Bromide 150 mg Oral Tablet: Methylnaltrexone Bromide 150 mg Oral Tablet
- Methylnaltrexone Subcutaneous Injection: Methylnaltrexone 12mg subcutaneous injection
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Methylnaltrexone Bromide 12 MG/0.6 ML Subcutaneous Solution [RELISTOR]_#1: Methylnaltrexone Bromide 12 MG Subcutaneous Solution
- Naloxegol Oral Tablets: Naloxegol oral tablets (total 25 mg)
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Naloxegol 25 MG Oral Tablet: Naloxegol 25 MG Oral Tablet
Period: Overall Study
Arm/Group | Methylnaltrexone Oral Tablets | Methylnaltrexone Subcutaneous Injection | Naloxegol Oral Tablets
Started | 4 | 3 | 5
Completed | 4 | 3 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Methylnaltrexone Oral Tablets: Methylnaltrexone oral tablets (total 450 mg) + subcutaneous water injection
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Methylnaltrexone Bromide 150 mg Oral Tablet: Methylnaltrexone Bromide 150 mg Oral Tablet
- Methylnaltrexone Subcutaneous Injection: Methylnaltrexone 12mg subcutaneous injection + sugar placebo tablet
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Methylnaltrexone Bromide 12 MG/0.6 ML Subcutaneous Solution [RELISTOR]_#1: Methylnaltrexone Bromide 12 MG Subcutaneous Solution
- Naloxegol Oral Tablets: Naloxegol oral tablets (total 25 mg) + subcutaneous water injection
  Eligible patients with complaint of opioid-induced constipation will receive this treatment after study enrollment. Time to bowel movement will be recorded until 3 hours in the emergency department, and patient will be contacted after 24 hours if bowel movement was not achieved after the 3 hours.
  Naloxegol 25 MG Oral Tablet: Naloxegol 25 MG Oral Tablet
- Total: Total of all reporting groups
Arm/Group | Methylnaltrexone Oral Tablets | Methylnaltrexone Subcutaneous Injection | Naloxegol Oral Tablets | Total
Number analyzed (Participants) | 4 | 3 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (28.3) | 55.3 (16.5) | 62.8 (18.8) | 57.8 (20.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 4 | 1 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 5 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Bowl Movement
Description: The primary outcome of this study is to determine the effectiveness of peripherally acting mu-opioid receptor antagonist therapy for patients presenting to the emergency department (ED) with opioid-induced constipation.
Time Frame: 24 hours
Population: The number of participants who had a successful bowl movement within 24 hours of administration of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Methylnaltrexone Oral Tablets | Methylnaltrexone Subcutaneous Injection | Naloxegol Oral Tablets
Number analyzed (Participants) | 4 | 3 | 5
Participants | 2 | 2 | 5

2. Secondary Outcome: Time to Bowl Movement Within 24 Hours
Description: The secondary outcome of this study is the time to effectiveness of subcutaneous versus oral therapy.
Time Frame: 24 hours after administration of study drug
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Methylnaltrexone Oral Tablets | Methylnaltrexone Subcutaneous Injection | Naloxegol Oral Tablets
Number analyzed (Participants) | 4 | 3 | 5
minutes | 292.5 (385.4) | 256.5 (21.9) | 270.2 (187.5)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Methylnaltrexone Oral Tablets | Methylnaltrexone Subcutaneous Injection | Naloxegol Oral Tablets
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 1/4 | 3/3 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylnaltrexone Oral Tablets (N=4) | Methylnaltrexone Subcutaneous Injection (N=3) | Naloxegol Oral Tablets (N=5)
Anxiety (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03523520/Prot_003.pdf
  • Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT03523520/SAP_005.pdf
  • Informed Consent Form (2020-04-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03523520/ICF_000.pdf